CLINICAL TRIAL: NCT04959760
Title: Clinical Evaluation of the BinaxNOW™ COVID-19 IgG Rapid Test Device and the BinaxNOW™ COVID-19 Antibody Self Test Clinical Study Protocol
Brief Title: BinaxNow COVID-19 IgG Rapid Test Device and Antibody Self Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Diagnostics Jena GmbH (Industry)
Responsible Party: Sponsor
Organization: Abbott Rapid Dx (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLDG-0511
Record Dates: First submitted 2021-07-01; First posted 2021-07-13 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Masking Description: Operator of the device will be blinded to the outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BinaxNow Covid-19 Antibody test (Experimental): The BinaxNOW™ Antibody Tests measure SARS-CoV-2 S-IgG antibodies.
  Interventions: Diagnostic Test: The BinaxNOW™ Antibody Tests measure IgG antibodies against SARS-CoV-2.

INTERVENTIONS:
Diagnostic Test: The BinaxNOW™ Antibody Tests measure IgG antibodies against SARS-CoV-2. — The BinaxNOW™ Antibody Tests measure IgG antibodies against SARS-CoV-2 in fingestick capillary blood and plasma samples.

SUMMARY:
Performance evaluation of the BinaxNOW™ COVID-19 IgG Rapid Test Device (Professional Use) and with BinaxNOW™ COVID-19 Antibody Self Test wehn used with fingerstick capillary whole blood and plasma samples. The BinaxNOW™ Antibody Tests are lateral flow tests that measure SARS-CoV-2 IgG antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 years of age or older.
2. Evaluable individuals with a prior confirmed SARS-CoV-2 infection with prior COVID-19 symptoms with symptoms onset > 14 days prior to the study, or symptoms onset 8-14 days prior to the study, or symptoms onset 0-7 days prior to study.OR

   Evaluable individuals confirmed negative by SARS-CoV-2 RT-PCR using a sample obtained within 7 days prior to or on the day of the study.
3. Participant agrees to complete all aspects of the study.

Exclusion Criteria:

1. Participant has already participated in this study on a previous occasion.
2. Participant is enrolled in a study to evaluate a new drug.
3. Participant has a visual impairment that cannot be restored using glasses or contact lenses.
4. Participant is unable or unwilling to provide informed consent.
5. Participant is a vulnerable person as deemed unfit for the study by the Principal Investigator.
6. Participant has a condition deemed unfit to safely perform the test by the investigator.
7. Participant is a practising health-care professional or laboratory scientist / technician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Clinical performance of the BinaxNOW™ COVID-19 IgG Rapid Test | Through study completion, an average of 6 months
  to evaluate the clinical performance of the BinaxNOW™ COVID-19 IgG Rapid Test Device when used by a professional user.
Clinical performance of the BinaxNOW™ COVID-19 Antibody Self-Test | Through study completion, an average of 6 months
  to evaluate the clinical performance of the BinaxNOW™ COVID-19 Antibody Self-Test when used by a lay person.

SECONDARY OUTCOMES:
Professional user usability | Through study completion, an average of 6 months
  Evaluation of the usability of the BinaxNOW™ COVID-19 IgG Rapid Test Device when used by a Professional User
Self Test user usability | Through study completion, an average of 6 months
  Evaluation of the usability of the BinaxNOW™ COVID-19 Antibody Self-Test when used by a lay person.
Matrix Equivalence Professional Use | Through study completion, an average of 6 months
  Validation of the Matrix Equivalence between the Fingerstick Whole Blood and Plasma samples when used with the BinaxNOW COVID-19 IgG Rapid Test Device.
Diagnostic sensitivity and specificity | Through study completion, an average of 6 months
  To determine the diagnostic sensitivity, specificity and overall agreement of the BinaxNOW™ COVID-19 Antibody Self Test as performed by lay users in comparison with the BinaxNOW™ COVID-19 IgG Rapid Test Device as performed by professional user.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Kordowich, Study Director — Abbott
Locations (5):
- United States (5):
  - Rush University Medical Center, Chicago, Illinois
  - Duke University Health System, Durham, North Carolina
  - Urgent Care Clinical Trials, Powdersville, South Carolina
  - Urgent Care Clinical Trials at Complete Health Partners, Nashville, Tennessee
  - Urgent Care Clinical Trials, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No